CLINICAL TRIAL: NCT00860132
Title: Economic Aspects Associated With the Implementation of an Orthogeriatric Setting in a General Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Abraham Adunsky, Director, Dept of Geriatric med & rehab, Sheba Medical Center
Other Study IDs: SHEBA-09-6962-AA-CTIL
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Hip Fracture
Keywords: hip fracture elderly orthogeriatric; cost effectiveness of hip fracture patients
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: a group of consecutive hip fracture patients admitted to a dedicated comprehensive orthogeriatric ward and a group of similar patients admitted to an orthopedic ward and later on transferred to geriatric rehab center

SUMMARY:
The economic and social burden of hip fractures is expected to increase dramatically, but financial resources remain limited. This calls for the investigation of innovative new forms of organization and integration of medical, surgical and rehabilitation services for these patients.

The study will investigate economical aspects associated with implementation of a comprehensive orthogeriatric ward for elderly hip fracture patients in a general hospital, compared with the classic model of orthopedic treatment followed by rehabilitation period.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture

Exclusion Criteria:

* Patients admitted for elective hip surgery
* Patients with multi-trauma injuries

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: approx 1000 patients admitted with traumatic hip fracture to an orthogeriatric ward, compared with approximately 1000 admissions to orthopaedic ward
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
cost-effectiveness | 1999-2007